CLINICAL TRIAL: NCT02780245
Title: Tranexamic Acid Versus Novel Uterine Cooling Technique in Reducing Blood Loss and Incidence of Postpartum Hemorrhage at Caesarean Section
Brief Title: Role of Tranexamic Acid Versus Uterine Cooling at Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Talkha Central Hospital (Other Government)
Responsible Party: Principal Investigator, Amro Mohamed Ibrahim Ibrahim Hetta, Dr. Amro M. Hetta, Talkha Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OG2
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Hemorrhage of Cesarean Section and/or Perineal Wound; Postpartum Hemorrhage; Uterine Atony
Keywords: Caesarean Section; Tranexamic Acid; Postpartum Hemorrhage; Ecbolics
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group (X) Prophylactic Tranexamic Acid (Experimental): Intravenously at 20 minutes preoperatively had an intervention of a single bolus TXA dose of 20•0 mg/kg, which was administered in Z solution (500•0 ml normal saline containing a prophylactic antibiotic 1•0 g) (NCT02739815).
  Interventions: Drug: Tranexamic Acid
- Group (Y) Intraoperative Uterine Cooling (Experimental): Firstly intravenously at 20 minutes preoperatively had only the Z solution, and secondly [Intraoperatively immediately following delivery of the fetus the uterus was been externalized in the usual fashion, and the body of the uterus cephalad to the hysterotomy incision was been wrapped in sterile surgical towels saturated in sterile and iced normal saline. These towels came from a sterile cooling pot set to 30 degrees Fahrenheit. Iced saline-soaked towels was been kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen].
  Interventions: Procedure: Intraoperative Uterine Cooling

INTERVENTIONS:
Drug: Tranexamic Acid — At 20 minutes preoperatively, TXA of 20 mg/kg was administered in Z Solution (500•0 ml normal saline containing a prophylactic antibiotic 1•0 g).
  Other Names: TXA
  Arms: Group (X) Prophylactic Tranexamic Acid
Procedure: Intraoperative Uterine Cooling — Intraoperatively immediately following delivery of the fetus the uterus was been externalized in the usual fashion, and the body of the uterus cephalad to the hysterotomy incision was been wrapped in sterile surgical towels saturated in sterile and iced normal saline. These towels came from a sterile cooling pot set to 30 degrees Fahrenheit. Iced saline-soaked towels was been kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen.
  Arms: Group (Y) Intraoperative Uterine Cooling

SUMMARY:
This study aims to compare role of a prophylactic predefined intravenous Tranexamic Acid dose versus intraoperative Uterine Cooling in reducing blood loss and incidence of postpartum hemorrhage at secondary CS.

DETAILED DESCRIPTION:
Bleeding during vaginal or operative delivery is always of prime concern. Despite significant progress in obstetric care 125,000 women die from obstetric hemorrhage annually in the world.

The incidence of CS is increasing, and the average blood loss during CS (1000 mL) is double the amount lost during vaginal delivery (500 mL). CS rate as high as 25-30% in many areas of the world. In Egypt the CS rate is 27.6 %, in United States of America, from 1970-2009 the CS rate rose from 4.5-32.9%, and declined to 32.8% of all deliveries at 2010. In spite of the various measures to prevent blood loss during and after CS, post-partum hemorrhage (PPH) continues to be the most common complication seen in almost 20% of the cases, and causes approximately 25% of maternal deaths worldwide, leading to increased maternal morbidity and mortality. Women who undergo a CS are much more likely to be delivered by a repeat operation in subsequent pregnancies. For women undergoing subsequent CS, the maternal risks are even greater like massive obstetric hemorrhage, hysterectomy, admission to an intensive care unit, or maternal death. Medications, such as oxytocin, misoprostol and prostaglandin F2α, have been used to control bleeding postoperatively.

TXA is a synthetic analog of the amino acid lysine, as an antifibrinolytic agent. Its intravenous administration has been routinely used for many years to reduce or prevent excessive hemorrhage in various medical conditions or disorders (helping hemostasis), also during and after surgical procedures like benign hysterectomy, open heart surgeries, scoliosis surgery, oral surgery, liver surgeries, total hip or knee arthroplasty, and urology. It has been shown to be very useful and efficient in reducing blood loss and incidence of blood transfusion in these surgeries, and decreases the risk of death in bleeding trauma patients. It was also included in the World Health Organization (WHO) Model List of Essential Medicines.

About its role in CS, some recent studies showed that TXA has advantage and useful effect safely in reducing blood loss and requirement of additional ecbolics. Its doses used intravenously to reduce blood loss at CS were a bolus of 1gm, 10 mg/kg , or 15 mg/kg which had an advantage over 10 mg/kg in anemic parturients.

A recent study by Mitchell et al. concluded that Uterine cooling during cesarean delivery was efficient enough to decrease blood loss and the incidence of postpartum hemorrhage.

This study aims to compare role of a prophylactic predefined intravenous Tranexamic Acid dose versus intraoperative Uterine Cooling in reducing blood loss and incidence of postpartum hemorrhage at secondary CS.

ELIGIBILITY:
Inclusion Criteria:

* Women who attended Talkha Central Hospital for planned or emergency secondary CS.
* Singleton pregnancy at term with gestational age (G.A) between 38±5 and 40 weeks.

Exclusion Criteria:

* Preoperative exclusion criteria were women who had any disorders of heart, liver, kidney, brain or blood, Abruptio placenta, placental abnormalities or accrete syndromes, Polyhydramnios, macrosomia, preeclampsia, allergy to TXA, history of thromboembolic disorders, or severe anemia.
* Intraoperative exclusion criteria was inability to exteriorize the uterus during CS for group (Y).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Total blood loss volume | Up to 3 hours
  Estimation of Total Blood Loss Volume (ml) during CS and in the PACU.

SECONDARY OUTCOMES:
Hematocrit value (Hct) | 6 hours postoperative period
  Estimating change in Pre- versus Post-operative hematocrit values (%) at 6 hours postoperatively.
Overall blood loss volume greater than 1000 cc | Up to 9 hours
  Estimation of overall blood loss volume during CS and up to 6 hours postoperatively
Need for Additional Ecbolics | Intraoperative
  Need for additional ecbolics to arrest and manage bleeding if there is a uterine atony
Need for other surgical measures to stop bleeding | Intraoperative
  Need for other surgical measures to stop bleeding (B-lynch denoting uterine atony, uterine artery ligation, hysterectomy)
Transfusion of Blood or Blood Products | Up to 3 hours
  Need for transfusion of blood or blood products during CS and in the PACU

OTHER OUTCOMES:
Blood Pressure | Up to 3 hours
  Measuring maternal blood pressure (mmHg) immediately postoperative and after 3 hours postoperative.
Maternal Side effects of intervention administered | Up to 9 hours
  Recording any Maternal side effects of interventions administered
APGAR Scores | up to 2 hours
  Recording of APGAR Score (/10) for all neonates immediately after delivery
Pulse Rate | Up to 3 hours
  Measuring maternal pulse rate (/minute) immediately postoperative and after 3 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Amro M Hetta, M.B., Ch.B., Principal Investigator — Talkha Central Hospital
Locations (1):
- Talkha Central Hospital, Al Mansurah, Al-Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarabrin O, Kaminskiy V, Galich S, Tkachenko R, Gulyaev A, Shcherbakov S, et al. Efficacy of tranexamic acid in decreasing blood loss during cesarean section. Critical Care 2012, 16(1): 1-189.
- [Background] Ahmed MR, Sayed Ahmed WA, Madny EH, Arafa AM, Said MM. Efficacy of tranexamic acid in decreasing blood loss in elective caesarean delivery. J Matern Fetal Neonatal Med. 2015 Jun;28(9):1014-8. doi: 10.3109/14767058.2014.941283. Epub 2014 Jul 28. PMID 25068947
- [Background] Gibbons L, Belizán JM, Lauer JA, Betrán AP, Merialdi M, Althabe F. The global numbers and costs of additionally needed and unnecessary caesarean sections performed per year: overuse as a barrier to universal coverage. World health report 2010, 30: 1-31.
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Wilson EC, Mathews TJ. Births: final data for 2010. Natl Vital Stat Rep. 2012 Aug 28;61(1):1-72. PMID 24974589
- [Background] Mayur G, Purvi P, Ashoo G, Pankaj D. Efficacy of tranexamic acid in decreasing blood loss during and after cesarean section: a randomized case controlled prospective study. J Obstet Gynecol India 2007, 57(3): 4.
- [Background] WHO Recommendations for the Prevention and Treatment of Postpartum Haemorrhage. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131942/ PMID 23586122
- [Background] Cahill AG, Stamilio DM, Odibo AO, Peipert JF, Ratcliffe SJ, Stevens EJ, Sammel MD, Macones GA. Is vaginal birth after cesarean (VBAC) or elective repeat cesarean safer in women with a prior vaginal delivery? Am J Obstet Gynecol. 2006 Oct;195(4):1143-7. doi: 10.1016/j.ajog.2006.06.045. Epub 2006 Jul 17. PMID 16846571
- [Background] Marshall NE, Fu R, Guise JM. Impact of multiple cesarean deliveries on maternal morbidity: a systematic review. Am J Obstet Gynecol. 2011 Sep;205(3):262.e1-8. doi: 10.1016/j.ajog.2011.06.035. Epub 2011 Jun 15. PMID 22071057
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- [Background] Shahid A, Khan A. Tranexamic acid in decreasing blood loss during and after caesarean section. J Coll Physicians Surg Pak. 2013 Jul;23(7):459-62. PMID 23823946
- [Background] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Background] Gaines-Dillard N, Bartley MK, Rosini JM. Tranexamic acid in the trauma patient. Nursing. 2016 Feb;46(2):60-2. doi: 10.1097/01.NURSE.0000476234.78599.e2. No abstract available. PMID 26760392
- [Background] Yehia AH, Koleib MH, Abdelazim IA, Atik A. Tranexamic acid reduces blood loss during and after cesarean section: A double blinded, randomized, controlled trial. Asian Pacific Journal of Reproduction 2014, 3(1): 53-56.
- [Background] Topsoee MF, Bergholt T, Ravn P, Schouenborg L, Moeller C, Ottesen B, Settnes A. Anti-hemorrhagic effect of prophylactic tranexamic acid in benign hysterectomy-a double-blinded randomized placebo-controlled trial. Am J Obstet Gynecol. 2016 Jul;215(1):72.e1-8. doi: 10.1016/j.ajog.2016.01.184. Epub 2016 Jan 30. PMID 26829509
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Movafegh A, Eslamian L, Dorabadi A. Effect of intravenous tranexamic acid administration on blood loss during and after cesarean delivery. Int J Gynaecol Obstet. 2011 Dec;115(3):224-6. doi: 10.1016/j.ijgo.2011.07.015. Epub 2011 Aug 27. PMID 21872857
- [Background] Sujata N, Tobin R, Kaur R, Aneja A, Khanna M, Hanjoora VM. Randomized controlled trial of tranexamic acid among parturients at increased risk for postpartum hemorrhage undergoing cesarean delivery. Int J Gynaecol Obstet. 2016 Jun;133(3):312-5. doi: 10.1016/j.ijgo.2015.09.032. Epub 2016 Feb 16. PMID 26952346
- [Background] Maged AM, Helal OM, Elsherbini MM, Eid MM, Elkomy RO, Dahab S, Elsissy MH. A randomized placebo-controlled trial of preoperative tranexamic acid among women undergoing elective cesarean delivery. Int J Gynaecol Obstet. 2015 Dec;131(3):265-8. doi: 10.1016/j.ijgo.2015.05.027. Epub 2015 Aug 15. PMID 26341174
- [Background] Wang HY, Hong SK, Duan Y, Yin HM. Tranexamic acid and blood loss during and after cesarean section: a meta-analysis. J Perinatol. 2015 Oct;35(10):818-25. doi: 10.1038/jp.2015.93. Epub 2015 Jul 30. PMID 26226243
- [Background] Simonazzi G, Bisulli M, Saccone G, Moro E, Marshall A, Berghella V. Tranexamic acid for preventing postpartum blood loss after cesarean delivery: a systematic review and meta-analysis of randomized controlled trials. Acta Obstet Gynecol Scand. 2016 Jan;95(1):28-37. doi: 10.1111/aogs.12798. Epub 2015 Nov 12. PMID 26698831
- [Background] Gupta A, Dwivedi Y, Shakya V, Srivastva U, Saxena A, Agarwal AM, et al. Efficacy of Tranexamic Acid in Reducing Perioperative Blood Loss During Caesarean Section: A Placebo Controlled Double Blind Study. International Journal of Scientific Research 2016, 5(3).
- [Background] Gungorduk K, Yildirim G, Asicioglu O, Gungorduk OC, Sudolmus S, Ark C. Efficacy of intravenous tranexamic acid in reducing blood loss after elective cesarean section: a prospective, randomized, double-blind, placebo-controlled study. Am J Perinatol. 2011 Mar;28(3):233-40. doi: 10.1055/s-0030-1268238. Epub 2010 Oct 26. PMID 20979013
- [Background] Goswami U, Sarangi S, Gupta S, Babbar S. Comparative evaluation of two doses of tranexamic acid used prophylactically in anemic parturients for lower segment cesarean section: A double-blind randomized case control prospective trial. Saudi J Anaesth. 2013 Oct;7(4):427-31. doi: 10.4103/1658-354X.121077. PMID 24348295
- [Background] Gai MY, Wu LF, Su QF, Tatsumoto K. Clinical observation of blood loss reduced by tranexamic acid during and after caesarian section: a multi-center, randomized trial. Eur J Obstet Gynecol Reprod Biol. 2004 Feb 10;112(2):154-7. doi: 10.1016/s0301-2115(03)00287-2. PMID 14746950
- [Background] Sekhavat L, Tabatabaii A, Dalili M, Farajkhoda T, Tafti AD. Efficacy of tranexamic acid in reducing blood loss after cesarean section. J Matern Fetal Neonatal Med. 2009 Jan;22(1):72-5. doi: 10.1080/14767050802353580. PMID 19165682
- [Background] Mitchell JL, Stecher J, Crowson J, Rich D. Uterine Cooling During Cesarean Delivery to Reduce Blood Loss and Incidence of Postpartum Hemorrhage: A Randomized Controlled Trial [31]. Obstetrics & Gynecology. 2015 May 1;125:9S-10S.